CLINICAL TRIAL: NCT05935150
Title: Omission of Sentinel Lymph Node Biopsy (SLNB ) in Early Breast Cancer Patients with Clinically Assessed Negative Axillary Lymph Nodes (cN0): a Phase II, Prospective Clinical Trial
Brief Title: Omission of SLNB in CN0 Early Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jue Wang, Prof., The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMSLNB
Record Dates: First submitted 2023-06-02; First posted 2023-07-07 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Clinically Assessed Negative Axillary Lymph Nodes; Sentinel Lymph Node
Keywords: breast cancer; clinically assessed negative axillary lymph nodes; sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OMSLNB (Experimental)
  Interventions: Procedure: Omit SLNB

INTERVENTIONS:
Procedure: Omit SLNB — All patients enrolled have to receive two or more imaging tests including axillary ultrasound assessed as axillary lymph node negative, and other tests including MRI, PET-CT, [18F]-FDG PET-MRI, axillary surgery will be omitted for eligible patients, and BCS or mastectomy (allowing breast reconstruction) will be chosen voluntarily by the patient under the premise of ensuring therapeutic efficacy, patients receiving BCS must undergo whole breast irradiation (WBI) after surgery, and the radiotherapy target area does not include the axillary region.

SUMMARY:
The OMSLNB trial adopts a prospective, single-arm, non-inferiority, phase-II, open-label study design. Patients with unilateral invasive breast cancer （tumor ≤3cm） and assessed as cN0 will be eligible for inclusion, enrolled patients are required to complete 2 or more imaging tests including axillary ultrasound assessed as axillary lymph node negative, and other tests including MRI, PET-CT, [18F]-FDG PET-MRI, eligible patients will avoid axillary surgery but will undergo breast surgery, which is not limited to breast-conserving surgery (BCS). So as to decrease the edema of upper arm, and finally improve the quality of life of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years;
2. Pathologically confirmed invasive breast cancer (regardless of pathological type) with a tumor diameter ≤ 3 cm, and planning to undergo breast surgery;
3. Negative axillary lymph nodes assessed by physical examination and imaging (2 or more of the following tests including ultrasound, breast MRI, breast PET-CT, breast PET-MRI, breast PET);
4. All patients are required to undergo immunohistochemical staining for Estrogen Receptor (ER), Progesterone Receptor (PR), human epidermal growth factor receptor 2 (HER2), Ki-67 proliferation index, and further fluorescence in situ hybridization (FISH) should be performed in HER2 2+ cases;
5. Good compliance, normal comprehension and ability to receive treatment and follow-up as required;
6. ECOG score 0-1;
7. Patients volunteered for this study and signed the informed consent form.

Exclusion Criteria:

1. Bilateral/lactating/pregnant breast cancer;
2. Previous history of malignant tumor or neoplasm;
3. Clinical or imaging confirmation of distant metastasis;
4. History of previous surgery on the affected axilla; or history of surgery affecting the function of the upper extremity;
5. Prior history of radiotherapy to the breast or chest;
6. Positive pathological margins after breast-conserving surgery or mastectomy;
7. Severe coagulation disorder, or a serious systemic disease, or an uncontrollable infection;
8. Aspartate aminortransferse (AST) and Alanine aminotransferase (ALT) ≥ 1.5 times the upper limit of normal, alkaline phosphatase ≥ 2.5 times the upper limit of normal, total bilirubin ≥ 1.5 times the upper limit of normal, serum creatinine ≥ 1.5 times the upper limit of normal; left ventricular injection fraction (LVEF) < 50% on cardiac ultrasound;
9. Inability to complete the full course of follow-up adjuvant therapy as prescribed by the doctor for various reasons;
10. No personal freedom and independent civil capacity;
11. Presence of mental disorders, addictions, etc;
12. Not eligible for enrollmentas as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
invasive Disease-Free Survival (iDFS) | 3 years
  Time interval from the surgery to invasive local-regional recurrence, distant metastasis, contralateral invasive breast cancer, or death from any cause.

SECONDARY OUTCOMES:
Breast cancer-related lymphoedema (BCRL) | 3 years
  Objective evaluation of breast cancer-related lymphoedema (BCRL) by arm circumference measurements and bioelectrical impedance technology. In our study, BCRL is diagnosed in two ways：① Relative Volume Change (RVC ) >10% in the affected upper extremity. ②Bioelectrical impedance technology: the impedance ratio is defined as the ratio of the impedance of the healthy upper limb to the impedance of the affected upper limb, and BCRL is diagnosed when the patient's impedance ratio is higher than the mean + 2 standard deviations (SD) of healthy controls, and BCRL will be diagnosed by meeting one of them.
Patient-reported outcomes (PROs) | 3 years
  Patients will be followed up with questionnaires using the FACT-B (Version 4.0) and Quick DASH at baseline, 1 week, 1, 3, 6, 12, 18, 24, and 36 months postoperatively, and the FACT-B scale will be used to assess changes in QoL from baseline to 3 years after surgery, and the Quick DASH scale will be used to assess changes in arm morbidity from baseline to 3 years after surgery.
Locoregional Recurrence (LRR) | 3 years
  This includes both local and regional recurrences. Local recurrence is defined as recurrence in the ipsilateral breast, chest wall, skin or surgical scar. Regional recurrence is defined as recurrence in the affected lymphatic drainage area, including the axilla, supraclavicular region, subclavicular region, and internal mammary node area.
Local Recurrence (LR) | 3 years
  Local recurrence is defined as recurrence in the ipsilateral breast, chest wall, skin or surgical scar.
Regional Recurrence (RR) | 3 years
  Regional recurrence is defined as recurrence in the affected lymphatic drainage area, including the axilla, supraclavicular region, subclavicular region, and internal mammary node area.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Zha, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Wang L, Wang Y, Ma L, Zheng R, Ding J, Gong Y, Yao H, Wang J, Zha X. Omission of sentinel lymph node biopsy in patients with clinically axillary lymph node-negative early breast cancer (OMSLNB): protocol for a prospective, non-inferiority, single-arm, phase II clinical trial in China. BMJ Open. 2024 Sep 10;14(9):e087700. doi: 10.1136/bmjopen-2024-087700. PMID 39260835